CLINICAL TRIAL: NCT05814822
Title: Targeting Insomnia to Improve Outcomes in Adults With Problematic Cannabis Use
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, J. Todd Arnedt, Professor of Psychiatry, Professor of Neurology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: HUM00222302; R01DA057297 (NIH)
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: Cannabis
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Marijuana Abuse | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Behavioral Therapy for insomnia (CBTi-CB-TM) (Experimental): Delivered via telemedicine
  Interventions: Behavioral: Cognitive Behavioral Therapy for insomnia (CBTi-CB-TM)
- Sleep Hygiene Education (Active Comparator): Delivered via telemedicine
  Interventions: Behavioral: Sleep Hygiene Education (SHE-TM)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for insomnia (CBTi-CB-TM) — Participants randomized to CBTi-CB-TM will participate in 6 individual telemedicine sessions delivered by a trained therapist to learn cognitive and behavioral strategies for insomnia.
  Arms: Cognitive Behavioral Therapy for insomnia (CBTi-CB-TM)
Behavioral: Sleep Hygiene Education (SHE-TM) — Participants randomized to SHE-TM will participate in 6 individual telemedicine sessions delivered by a trained therapist to learn sleep hygiene and educational strategies for insomnia.
  Arms: Sleep Hygiene Education

SUMMARY:
This study will compare the efficacy of telemedicine-delivered cognitive behavioral therapy for insomnia tailored for people using cannabis for sleep (CBTi-CB-TM) to telemedicine-delivered sleep hygiene education (SHE-TM) on sleep, cannabis use, and daytime functioning. We will also evaluate the effects of CBTi-CB-TM on fundamental sleep regulatory system - homeostatic sleep drive - and its association with clinical outcomes.

ELIGIBILITY:
INCLUSION CRITERIA

* 21 years of age and older, the age needed to obtain full legal access to cannabis in Michigan
* Self-reported chronic insomnia (nighttime symptoms of difficulty initiating and/or maintaining sleep and/or early morning awakenings on ≥3 nights for ≥3 months with daytime impairment), consistent with DSM-5 diagnosis of Insomnia Disorder
* Insomnia Severity Index (ISI) score ≥11, indicative of at least "mild" insomnia
* A positive urine drug screen (UDS) for cannabis33
* Self-reported use of cannabis at least three times weekly for the past month
* Stable residence (e.g., stable sleep arrangements), consistent access to Wi-Fi, and ability to travel to Ann Arbor for sleep laboratory assessments

EXCLUSION CRITERIA

* Individuals who do not understand English (read and spoken)
* Individuals judged unable to provide informed consent (e.g., intoxication, mental incompetence)
* Diagnosis or high suspicion of a sleep disorder other than insomnia
* Lifetime diagnosis of psychotic disorder or bipolar disorder; current post-traumatic stress disorder that directly interferes with sleep
* Terminal or progressive physical illness (e.g., cancer) or neurological degenerative disease (e.g., dementia)
* Use of medications known to have initiated their insomnia (e.g., steroids)
* Previous receipt of CBTi
* Self-reported pregnancy
* Self-reported regular work schedule of rotating or night (3rd) shift work
* Other conditions and situations, medical or otherwise, that preclude meaningful and/or safe participation in CNT/SHE and study procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of cannabis use as measured by the Timeline Followback (TLFB) | Up to 6 months after intervention, approximately 32 weeks
  Changes in frequency of cannabis use will be evaluated over the past 30 days using the Timeline Followback, widely considered the "gold standard" tool for assessing daily substance use. It will be used to measure the frequency of use of THC-containing cannabis products used across all modalities guided by pictorial aids. Participants are asked to specify motivations behind cannabis use, including recreation, medicinal use, sleep aid, or other reasons. We will collect data on alcohol and other substance use during the interview. The primary outcome is frequency of cannabis use per day across all modalities. Participants obtain cannabis from a variety of sources and thus dose assessments using retrospective recall would not be reliable. We therefore chose frequency as our primary outcome, which is also recommended by expert consensus.
Insomnia Severity Index (ISI) total score measured by the Insomnia Severity Index (ISI) | Up to 6 months after intervention, approximately 32 weeks
  Changes in insomnia severity from baseline to post-treatment is assessed with the 7-item Insomnia Severity Index (ISI), a self-administered assessment of global insomnia severity over the past 2 weeks that ranges in score from 0 to 28, with higher scores indicating more severe insomnia symptoms (0-7 no clinical insomnia, 8-14 mild insomnia severity, 15-22 moderate insomnia severity, 23-28 severe insomnia severity). The primary outcome is ISI total score.
Mental Composite Score (MCS-12) as assessed by the 12-item Short-Form Health Survey (SF-12) | Up to 6 months after intervention, approximately 32 weeks
  The 12-item Short-Form Health Survey (SF-12) is a short-form quality of life measure derived from the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). The primary outcome is the Mental Component Summary Score (MCS-12), which ranges from 0-100, with higher scores indicating better health

SECONDARY OUTCOMES:
EEG Delta Activity | Pre- and Post-Intervention
  The outcome of interest is change in the rate of dissipation of Non-Rapid Eye Movement (NREM) sleep Slow Wave Activity (SWA) over the course of the night (measured with the best-fit slope based on exponential regressions), but we will additionally evaluate change in SWA power in the first NREM period and averaged across the night

CONTACTS AND LOCATIONS:
Overall Officials: Todd Arnedt, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No